CLINICAL TRIAL: NCT01806649
Title: A Phase II Study of BKM120; a Pan-PI3K Inhibitor in Patients With Esophageal Squamous Cell Carcinoma After Failure of First Line Chemotherapy
Brief Title: BKM120 in Esophageal Squamous Cell Carcinoma After Failure of First Line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated to continue any clinical trials with study drug
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Arunee Dechaphunkul, Dr, Prince of Songkla University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 551691411
Record Dates: First submitted 2013-03-01; First posted 2013-03-07 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; second line therapy; BKM120
MeSH Terms: conditions — Esophageal Neoplasms | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 (Experimental): BKM120, starting at 100 mg oral once daily
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120

SUMMARY:
There is a need for more effective therapy for patients with esophageal squamous cell carcinoma who developed disease progression after first line therapy. Currently, there is no standard second-line therapy for this disease.

BKM-120 is a pan-PI3K inhibitor currently tested in clinical trials. In a cellular model of oral-esophageal carcinogenesis, it has shown that EGFR overexpression activated PI3/AKT pathway. Therfore, there is interest to see the efficacy and safety of BKM120 in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided a signed Informed Consent Form (ICF) obtained prior to any screening procedure.
* Age ≥ 18 years old
* Histologically confirmed diagnosis of esophageal squamous cell carcinoma and available archival tissue for evaluation of further studies.
* Metastatic or unresectable disease
* Received one prior chemotherapy or biological therapy regimen for unresectable or metastatic disease
* More than 30 days since prior chemotherapy, surgery, radiotherapy, or investigational agents
* Measurable disease in at least 1 diameter by CT scan or MRI as per RECIST 1.1 criteria
* No evidence of brain metastasis
* ECOG ≤ 2
* Patient has adequate bone marrow and organ function

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin ≥ 9.0 g/dL
  * INR ≤ 2
  * Potassium, calcium, magnesium within normal limits for the institution
  * Serum Creatinine ≤ 1.5 x ULN or Creatinine clearance > 60 mL
  * AST and ALT not more than 2.5 times ULN (not more than 5.0 times ULN if there is liver metastasis)
  * Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
  * Fasting serum glucose < 1.5 times ULN

Exclusion Criteria:

* Patient has received previous treatment with PI3K inhibitors
* Patient has symptomatic CNS metastases
* Patients with controlled and asymptomatic CNS metastases may participate in this trial. As such, the patient must have completed any prior treatment for CNS metastases > 28 days (including radiotherapy and/or surgery) prior to enrollment in this study and should not be receiving chronic corticosteroid therapy for the CNS metastases.
* Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment, (with the exception of nonmelanoma skin cancer or cervical carcinoma in situ.
* Patient has any of the following mood disorders as judged by the Investigator or a Psychiatrist, or meets the cut-off score of ≥ 10 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts ideation in the PHQ-9 (independent of the total score of the PHQ-9)
* Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) ≥ CTCAE grade 3 anxiety
* Patient is concurrently using other approved or investigational antineoplastic agent
* Patient has had major surgery within 28 days prior to starting study drug or has not recovered from major side effects of the surgery
* Patient has poorly controlled diabetes mellitus(HbA1c > 8 %)
* Patient has active cardiac disease including any of the following:

  * LVEF < 50%
  * QTc > 480 msec on screening ECG (using the QTcF formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
* Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication
* Conduction abnormality requiring a pacemaker
* Valvular disease with documented compromise in cardiac function
* Symptomatic pericarditis
* Patient has a history of cardiac dysfunction including any of the following;

  * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
* Documented cardiomyopathy
* Patient is currently receiving treatment with QT prolonging medication known to have a risk to induce Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Inability to swallow, impaired gastrointestinal (GI) function, or GI disease that would significantly alter the absorption of study drugs or preclude the use of oral medications
* Patient has other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate her participation in the clinical study (e.g.,chronic pancreatitis, active chronic hepatitis etc.)
* Patient is currently being treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
disease control rate | 16 weeks
  16-week disease control rate using RECIST 1.1 criteria

SECONDARY OUTCOMES:
safety | each follow up visit, assessed up to 12 months
  Safety data will be assessed at each study visit using CTCAE version 4.0
progression-free survival | Time from day 1 to date of documented disease progression or death, assessed up to 12 months
overall survival | Time from day 1 to date of death, assessed up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Arunee Dechaphunkul, MD, Principal Investigator — Prince of Songkla University, Thailand
Locations (1):
- Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Background] Bendell JC, Rodon J, Burris HA, de Jonge M, Verweij J, Birle D, Demanse D, De Buck SS, Ru QC, Peters M, Goldbrunner M, Baselga J. Phase I, dose-escalation study of BKM120, an oral pan-Class I PI3K inhibitor, in patients with advanced solid tumors. J Clin Oncol. 2012 Jan 20;30(3):282-90. doi: 10.1200/JCO.2011.36.1360. Epub 2011 Dec 12. PMID 22162589
- [Background] Heeg S, Hirt N, Queisser A, Schmieg H, Thaler M, Kunert H, Quante M, Goessel G, von Werder A, Harder J, Beijersbergen R, Blum HE, Nakagawa H, Opitz OG. EGFR overexpression induces activation of telomerase via PI3K/AKT-mediated phosphorylation and transcriptional regulation through Hif1-alpha in a cellular model of oral-esophageal carcinogenesis. Cancer Sci. 2011 Feb;102(2):351-60. doi: 10.1111/j.1349-7006.2010.01796.x. Epub 2010 Dec 12. PMID 21156006